CLINICAL TRIAL: NCT04274192
Title: Effect of Synchronized vs. Continuous High Flow Nasal Cannula Using Neurally Adjusted Ventilatory Assist on Work of Breathing in Infants With Bronchopulmonary Dysplasia
Brief Title: Effect of Synchronized vs. Continuous HFNC Using NAVA on WOB in Infants With BPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left and study not feasible as written in the protocol
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 239863
Record Dates: First submitted 2019-08-29; First posted 2020-02-18 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Alternating between Synchronized and Continuous HFNC at 6 and 8 LPM (starting with synchronized) (Experimental): Subjects will first receive HFNC synchronized to his/her own efforts via NAVA at 6 LPM followed by continuous HFNC at 6 LPM and then HFNC synchronized to his/her own efforts via NAVA at 8 LPM followed by continuous HFNC at 8 LPM
  Interventions: Other: Synchronized HFNC at 6 liters per minute (LPM); Other: Continuous HFNC at 6 liters per minute (LPM); Other: Synchronized HFNC at 8 liters per minute (LPM); Other: Continuous HFNC at 8 liters per minute (LPM)
- Alternating between Synchronized and Continuous HFNC at 6 and 8 LPM (starting with continuous) (Active Comparator): Subjects will first receive continuous HFNC at 6 LPM followed by HFNC synchronized to his/her own efforts via NAVA at 6 LPM. Next, subjects will receive continuous HFNC at 8 LPM followed by HFNC synchronized to his/her own efforts via NAVA at 8 LPM.
  Interventions: Other: Synchronized HFNC at 6 liters per minute (LPM); Other: Continuous HFNC at 6 liters per minute (LPM); Other: Synchronized HFNC at 8 liters per minute (LPM); Other: Continuous HFNC at 8 liters per minute (LPM)

INTERVENTIONS:
Other: Synchronized HFNC at 6 liters per minute (LPM) — HFNC given in synchrony with the subject's own respiratory effort using NAVA at 6 LPM
Other: Continuous HFNC at 6 liters per minute (LPM) — Standard HFNC therapy at 6 LPM
Other: Synchronized HFNC at 8 liters per minute (LPM) — HFNC given in synchrony with the subject's own respiratory effort using NAVA at 8 LPM
Other: Continuous HFNC at 8 liters per minute (LPM) — Standard HFNC therapy at 8 LPM

SUMMARY:
Patients will be randomized to begin the study with either NAVA-synchronized or continuous HFNC. Each patient will receive two 15-minute trials at different levels of continuous HFNC and two 15-minute trials at corresponding levels of synchronized HFNC. In synchronized HFNC, using the NIV NAVA mode on the ventilator each subject will receive a constant minimum flow, but with each neurally triggered breath (as measured with an Edi catheter), an additional flow will be given to the patient. This differs from continuous HFNC in which the subject receives a constant flow without variation. Subjects will be observed during the entirety of these trials. Values for the primary and secondary outcomes will be monitored, recorded, and calculated.

DETAILED DESCRIPTION:
Prior to the study period each subject will have the following monitoring equipment placed (if not already present): Edi catheter, transcutaneous monitor (TCM4, Radiometer, Brea, CA, USA) to measure CO2 and O2 levels, pulse oximeter probe (MasimoSET, Irvine, CA, USA) to measure oxygen saturations and heart rate, and RIP bands (SleepSense, MFI Medical, San Diego, CA, USA) around the chest and abdomen to measure breathing movements and relative tidal volume.

Each subject will be randomized on the day the study is to occur to begin with either NAVA-synchronized or continuous HFNC before crossing over to the other mode to serve as his/her own control. The same RAM cannula will be used in both study arms and will provide a leak of 60-80% as recommended by the product manual. The delivery of high flow during both synchronized and continuous HFNC will be given at two commonly provided levels of high flow: 6 LPM and 8 LPM, given in the same order in each mode (6 LPM then 8 LPM). Each subject will receive 15-minute trials of each mode-level combination, for a total of four trials. During each trial, the first 10 minutes will be used for stabilization, and the last 5 minutes will be used for data collection, as has been done in previous trials. Thus, the mode-level combinations of the trials will be as follows: for infants randomized to begin with synchronized support: synchronized-6 LPM, synchronized-8 LPM, unsynchronized-6 LPM, unsynchronized-8 LPM. For infants randomized to begin with unsynchronized support: unsynchronized-6 LPM, unsynchronized-8 LPM, synchronized-6 LPM, unsynchronized-8 LPM.

The flows described in the NAVA-synchronized trials refer to the peak flow provided during inspiration. A baseline flow rate of 2 LPM will be provided expiration in these trials (using the PEEP setting corresponding to the appropriate flow rate). During the unsynchronized trials, the continuous high flow rate will be provided (as is common practice with the use of HFNC). During the NAVA-synchronized HFNC trials, the Edi trigger will be set to 0.5 microvolts, apnea time to 5 seconds, back up rate to 10 breaths per minute, and backup pressure settings will be set to provide an estimated peak flow of 6 or 8 LPM according to the designated trial (again, using the pressure setting corresponding to the appropriate flow rate).

During NAVA-synchronized HFNC, the NIV NAVA mode will be set in such a way that synchronized HFNC will be provided. A minimal end-expiratory flow of 2 LPM will be provided using the positive end expiratory pressure (PEEP) setting in the NIV NAVA mode on the ventilator. The PEEP setting corresponding to 2 LPM via the pneumotachograph will be used. In order to deliver the desired peak flow rate with each neurally-triggered breath, a NAVA level of 15 cmH2O/μV will be set, then the maximum pressure setting that corresponds to the desired flow rate using the pneumotachograph will be used for the study. The subject will thus be provided with "synchronized HFNC". This contrasts with the constant-flow trials when subjects will receive a constant and non-synchronized flow using the HFNC software on the ventilator.

Servo-u ventilators and Servo Tracker Software (Maquet Critical Care, Solna, Sweden) will be used in order to track Edi signal. The MP100 Biopac data acquisition (Biopac Systems Inc., Goleta, CA, USA) will be used to collect data from the monitoring devices. HFNC will be delivered using appropriately sized RAM cannula to allow for air leak around the subject's nares. Persistent bradycardia (less than 100 beats per minutes), desaturation (<85%), or hypercarbia (transcutaneous CO2 >70) will result in cessation of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age greater than 28 days
* Gestational age at birth less than 32 weeks and 6 days
* Diagnosis of BPD (supplemental oxygen requirement for greater than or equal to 28 days)
* Currently receiving noninvasive ventilation support (NIV NAVA, NIPPV, nCPAP, HFNC)

Exclusion Criteria:

* Major congenital anomalies of the heart and lungs
* Post menstrual age greater than 50 weeks 0 days
* Oxygen requirement greater than 40%

Ages: 28 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry E Courtney, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one participant was enrolled. The study was subsequently stopped.
  Reasons:
  1. Lengthy study recruitment pause due to COVID
  2. Principal investigator left the institution.
  3. Insufficient staff to revise protocol and continue study.
  4. Continuation of study would require significant protocol revision due to flow/pressure/ventilator interactions for this trial.
Groups:
- Synchronized HFNC First: Subjects will first receive HFNC synchronized to his/her own efforts via NAVA at 6 LPM followed by continuous HFNC at 6 LPM and then HFNC synchronized to his/her own efforts via NAVA at 8 LPM followed by continuous HFNC at 8 LPM
- Continuous HFNC First: Subjects will first receive continuous HFNC at 6 LPM followed by HFNC synchronized to his/her own efforts via NAVA at 6 LPM and then continuous HFNC at 8 LPM followed by HFNC synchronized to his/her own efforts via NAVA at 8 LPM.
Period: Overall Study
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Started | 1 | 0
Completed (Using the equipment available, we were unable to administer the 6 LPM (per the protocol), so this subject did not receive all of the interventions and therefore did not complete the study. We subsequently terminated the study due to lack of protocol feasibility and the departure of the original PI.) | 0 | 0
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Using the equipment available, we were unable to administer the 6 LPM (per the protocol), so this subject could not receive all of the interventions described in the protocol and therefore did not complete the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Synchronized HFNC First | Continuous HFNC First | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: days] | 56 [56 to 56] |  | 56 [56 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patient was caucasian.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 1 | 0 | 1
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Work of Breathing
Description: estimated using swing Edi
Time Frame: 15 minutes
Population: Only one patient was enrolled, but that subject did not complete the study due to a protocol violation related to a lack of protocol feasibility with the equipment available. Therefore, there are no outcome data.
Groups:
- Synchronized HFNC: This will be the experimental arm in which subjects will receive HFNC synchronized to his/her own efforts via NAVA
  Synchronized HFNC: HFNC given in synchrony with the subject's own respiratory effort using NAVA
  Continuous HFNC: Standard HFNC therapy
- Continuous HFNC: This arm will be considered the control arm in which subjects will receive continuous HFNC.
  Synchronized HFNC: HFNC given in synchrony with the subject's own respiratory effort using NAVA
  Continuous HFNC: Standard HFNC therapy
Arm/Group | Synchronized HFNC | Continuous HFNC
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Thoracoabdominal Asynchrony
Description: estimated by phase angle calculated by data obtained from respiratory inductance plethysmography bands
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Uncalibrated Tidal Volume
Description: as estimated using data from respiratory plethysmography bands
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: FiO2 Requirement
Description: the amount of oxygen patient requires during the study
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Oxygen Saturation
Description: measured by pulse oximetry
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Transcutaneous Oxygen Level
Description: using a transcutaneous oxygen monitor
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Transcutaneous Carbon Dioxide Level
Description: using a transcutaneous carbon dioxide monitor
Time Frame: 15 minutes
Population: as for outcome 1
Arm/Group | Synchronized HFNC First | Continuous HFNC First
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Until the end of the treatment, approximately 1 day per subject
Description: 0 subjects were enrolled in the "continuous HFNC" arm, therefore 0 were at risk for SAEs, All-cause mortality, or Other AEs
Arm/Group | Synchronized HFNC First | Continuous HFNC First
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synchronized HFNC First (N=1) | Continuous HFNC First (N=0)
Study team error (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Nothing adverse occurred and the event was a result of a safety precaution we were not aware of on the ventilator, which did not permit pressure recording low enough for 6LPM during the NAVA data collection.

LIMITATIONS AND CAVEATS:
Using the equipment available, we were unable to administer the 6 LPM (per the protocol), so this subject did not receive all of the interventions and therefore did not complete the study.

We subsequently terminated the study due to lack of protocol feasibility and the departure of the original PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT04274192/Prot_SAP_000.pdf